CLINICAL TRIAL: NCT02511769
Title: WEB MAP Intervention for Youth With Sickle Cell Disease
Brief Title: Web-MAP Intervention for Youth With Sickle Cell Disease
Acronym: Web-MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Head, Division of Pain and Palliative Medicine, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-032
Record Dates: First submitted 2014-09-25; First posted 2015-07-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WEB-MAP CBT (Experimental): Web-MAP Group. Participants will have access to the full version of the web program. They will be asked to log in to the website using their own personal computer at home, work, school, or a public library. Participants in the Web-MAP group will have access to treatment modules and daily diaries on the web site. The online treatment will take between 8 and 9 weeks for participants to complete. Children and parents will be asked to log onto the web site, read through the treatment modules, and complete practice assignments to learn new skills (e.g., relaxation). Adolescents and parents will be asked to complete a total of 8 modules each.
  Interventions: Behavioral: WEB-MAP CBT
- WEB-MAP Educational Control Group (Active Comparator): OPEC (Online Patient Education Control) Group: The purpose of the patient education control group is to control for time, attention, and computer usage. This group will serve as an attention control condition. Children will continue with the standard medical care that has been prescribed for their pain problem. Children and parents will be provided with access to a revised version of the Web-MAP study website, which will have two functional components: 1) information from publicly available educational websites about pediatric chronic pain management, 2) diary and assessments. This version of the website differs from the one accessed by the treatment condition in that it does not provide access to behavioral and cognitive skills training via treatment modules for children and parents.
  Interventions: Behavioral: WEB-MAP Educational Control Group

INTERVENTIONS:
Behavioral: WEB-MAP Educational Control Group — OPEC (Online Patient Education Control) Group: The purpose of the patient education control group is to control for time, attention, and computer usage. This group will serve as an attention control condition. Children will continue with the standard medical care that has been prescribed for their pain problem. Children and parents will be provided with access to a revised version of the Web-MAP study website, which will have two functional components: 1) information from publicly available educational websites about pediatric chronic pain management, 2) diary and assessments. This version of the website differs from the one accessed by the treatment condition in that it does not provide access to behavioral and cognitive skills training via treatment modules for children and parents.
  Arms: WEB-MAP Educational Control Group
Behavioral: WEB-MAP CBT — Web-MAP Group: Participants will have access to the full version of the web program. They will be asked to log in to the website using their own personal computer at home, work, school, or a public library. Participants in the Web-MAP group will have access to treatment modules and daily diaries on the web site. The online treatment will take between 8 and 9 weeks for participants to complete. Children and parents will be asked to log onto the web site, read through the treatment modules, and complete practice assignments to learn new skills (e.g., relaxation). Adolescents and parents will be asked to complete a total of 8 modules each.
  Arms: WEB-MAP CBT

SUMMARY:
The proposed study will determine whether the efficacy of WebMAP cognitive behavioral therapy (CBT) treatment study generalizes to pediatric sickle cell disease (SCD), and explore whether the intervention is feasible and acceptable to this population. Feasibility of multi-institutional recruitment from sickle cell centers will also be determined. The short-term goal is to produce preliminary data to apply for an R01 proposal to carry out a multi-institutional randomized controlled trial (RCT) of internet-delivered behavioral intervention in a large population of youth with SCD. The long-term goal of this research is to develop effective, easily accessible, behavioral pain interventions for youth with SCD to reduce the long-term impact of pain on function, quality of life, and health service use in this population.

The design of this study is an experimental 2 (group) x 3 (time of measurement) randomized controlled trial design to test the acceptability and efficacy of the Web-MAP intervention in reducing pain and functional impairment in youth with sickle cell disease. (Figure 1) Subjects will be randomized to either the behavioral intervention or the online patient education control group. The treatment protocol will be implemented over 8 weeks in Internet-based treatment modules. The primary study outcome is pain and functional impairment measured at baseline, immediately post-treatment, and at 3-month follow-up.

DETAILED DESCRIPTION:
The proposed study will determine whether the efficacy of WebMAP generalizes to pediatric SCD, and explore whether the intervention is feasible and acceptable to this population. Feasibility of multi-institutional recruitment from sickle cell centers will also be determined. The short-term goal is to produce preliminary data to apply for an R01 proposal to carry out a multi-institutional randomized controlled trial (RCT) of internet-delivered behavioral intervention in a large population of youth with SCD. The long-term goal of this research is to develop effective, easily accessible, behavioral pain interventions for youth with SCD to reduce the long-term impact of pain on function, quality of life, and health service use in this population.

The design of this study is an experimental 2 (group) x 3 (time of measurement) randomized controlled trial design to test the acceptability and efficacy of the Web-MAP intervention in reducing pain and functional impairment in youth with sickle cell disease. (Figure 1) Subjects will be randomized to either the behavioral intervention or the online patient education control group. The treatment protocol will be implemented over 8 weeks in Internet-based treatment modules. The primary study outcome is pain and functional impairment measured at baseline, immediately post-treatment, and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Documented sickle cell disease (verified by physician at SCD center if referred participant is a self referral)
* 11-18 years old
* Parental/patient consent and patient assent
* Internet and computer or smartphone access
* Score of >3 on the SCPBI-Y

Exclusion Criteria:

* Primary language spoken other than English
* 11<Age≤19
* Serious comorbid chronic condition (e.g., diabetes, arthritis, cancer)
* More than 4 sessions of outpatient behavioral therapy for pain management in the 6 months prior to the time of screening

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
Efficacy in pain reduction | 6 months
  We will compare pain intensity (pain scores), pain burden (Sickle Cell Pain Burden Interview), activity limitations (Child Activity Limitations Interview), quality of life (PedsQL), and health service use, and their corresponding changes from baseline to T2 (immediately after finishing the treatment arm) and T3 (6 months after enrollment in study). We will used a paired sample t-test.

SECONDARY OUTCOMES:
Efficacy of reducing depressive symptoms | 6 months
  We will compare changes changes in depressive symptoms using the Centers for Epidemiological Study Depression scale from baseline to T2 (immediately after finishing the treatment arm) and T3 (6 months after enrollment in study). We will used a paired sample t-test.

OTHER OUTCOMES:
Feasibility of WEB-MAP program | 6 months
  We will conduct interviews with participants of the study using a script to start a dialogue on how user friendly their interface is, perceived difficulties or barriers, improvements to make, and general overall feedback to modify the program.

CONTACTS AND LOCATIONS:
Overall Officials: William T Zempsky, MD, MPH, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- CCMC, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No